CLINICAL TRIAL: NCT04651647
Title: Is Open Bone Graft Always Necessary When Treating Subtrochanteric Nonunion With a Reamed Intramedullary Nail?
Brief Title: Bone Graft in Aseptic Subtrochanteric Nonunion
Status: Completed | Type: Observational
Sponsor: Jae Hoon Jang (Other)
Collaborators: Pusan National University Yangsan Hospital (Other)
Responsible Party: Sponsor-Investigator, Jae Hoon Jang, Associate Professor, Pusan National University Hospital
Organization: Pusan National University Hospital (Other)
Other Study IDs: realjang
Record Dates: First submitted 2020-11-20; First posted 2020-12-03 (Actual); Last update posted 2020-12-03 (Actual); Status verified 2020-11

CONDITIONS: Subtrochanteric Nonunion
Keywords: subtrochanteric nonunion; intramedullary nail; bone graft
MeSH Terms: interventions — Reoperation

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Bone graft group: The bone graft group (n=19) who underwent open nailing with open bone graft for aseptic subtrochanteric nonunion
  Interventions: Procedure: Revision surgery with / without open bone graft
- Non bone graft group: The non-BG group (n=18) who underwent closed reamed nailing without bone graft for aseptic subtrochanteric nonunion
  Interventions: Procedure: Revision surgery with / without open bone graft

INTERVENTIONS:
Procedure: Revision surgery with / without open bone graft — Removal of previous implant and re-alignment and re-fixation using intramedullary nail with (bone graft group) / without (non bone graft group) open bone graft

SUMMARY:
This study aimed to compare the radiologic results between closed nailing without bone graft (BG) and open nailing with BG for subtrochanteric nonunion and to determine when open BG should be considered.

DETAILED DESCRIPTION:
In this retrospective study, we investigated the patients who underwent surgical intervention for subtrochanteric nonunion between January 2008 and March 2018 in two institutions. The cases with infection, large bone defect, pathologic fracture, open fracture, previous surgery using plate, and follow-up less than 1 year were excluded. We compared the demographic details and radiologic results between patients who underwent the open procedure with BG (BG group) and the closed procedure without BG (non-BG group) as a historical control, and risk factors for the failure of revision surgery were evaluated.

ELIGIBILITY:
Inclusion Criteria:

* Patients who underwent surgical intervention using intramedullary nailing for aseptic subtrochanteric nonunion

Exclusion Criteria:

* The cases with infection, large bone defect, pathologic fracture, open fracture, previous and revision surgery using plate, and follow-up less than 1 year

Ages: 32 Years to 82 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients who visited our institutions for surgical treatment of subtrochanteric nonunion and underwent surgical intervention in the institutions.
Sampling Method: Probability Sample
Enrollment: 37 (Actual)
Dates: Start 2008-01-01 (Actual); Primary Completion 2018-03-31 (Actual); Study Completion 2019-11-01 (Actual)

PRIMARY OUTCOMES:
bony union | The time when bone union was achieved after surgery
  Union was defined as painless full weight bearing with the absence of fracture line or bridging callus across at least three cortices on the AP and lateral views.
risk factors for nonunion | One year after surgery
  Determining when open procedure with bone graft should be considered by analyzing risk factors for nonunion.

CONTACTS AND LOCATIONS:
Locations (1):
- Pusan National University Hospital, Busan, South Korea

IPD SHARING:
Plan to Share IPD: Undecided
I would like to determine whether or not to share IPD after publication.